CLINICAL TRIAL: NCT00767325
Title: Multi-Center, Open Label Study to Assess Early Response to Abatacept With Background Methotrexate Using Power Doppler Ultrasonography in Patients With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate
Brief Title: A Rheumatoid Arthritis Study to Assess Early Response to Abatacept+MTX as Defined by Improvement of Synovitis Measures by Power Doppler Ultrasonography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IM101-179
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abatacept, 10 mg/kg (Experimental)
  Interventions: Drug: Abatacept; Drug: Methotrexate

INTERVENTIONS:
Drug: Abatacept — Abatacept, 10 mg/kg, solution given intravenously on Days 1, 15, 29,57, 85, 113, 141, and 169
  Other Names: Orencia®; BMS-188667
Drug: Methotrexate — Methotrexate administered in a dose of 15 mg/week or higher for at least 3 months and at a stable dose for at least 28 days prior to baseline

SUMMARY:
The purpose of the study is to assess early signs of response to abatacept+methotrexate in metacarpophalangeal joints in both hands using power Doppler ultrasonography in patients with active rheumatoid arthritis.

ELIGIBILITY:
Key inclusion riteria:

* Disease activity defined by a disease activity score 28-C-reactive protein >3.2, or meeting the following criteria: a tender joint count ≥6; a swollen joint count ≥6; C-reactive protein measurement greater than the upper limit of normal
* Diagnosis of rheumatoid arthritis for longer than 6 months from time of initial diagnosis
* Total synovitis power Doppler ultrasonography (PDUS) score >1 for at least 2 metacarpophalangeal (MCP) joints (MCP2-5) and a total synovitis PDUS score ≥1 for at least 1 other MCP joint (MCP2-5)
* Concomitant treatment with methotrexate at a dose ≥15 mg for at least 3 months before Day 1 and a stable dose for the last 28 days before Day 1
* No treatment with any background nonbiologic disease-modifying antirheumatic drug (DMARD) other than methotrexate for at least 28 days before treatment (Day 1)
* Stable dose of corticosteroids equivalent of 10 mg prednisone /day during the 28 days prior to Day 1
* Naive to treatment with biologic DMARDs

Key exclusion criteria:

* Women of childbearing potential who are unwilling or unable to use birth control
* Women who are pregnant or breastfeeding
* Meeting all diagnostic criteria for any other rheumatic disease
* Previous MCP arthroplasty, with such a procedure scheduled, or anticipating the need for such a procedure during the study. Participants who had undergone or were scheduled to undergo joint arthroplasties other than of the MCP joints were permitted to enroll in the study provided all other eligibility criteria were met.
* Active vasculitis of a major organ system with the exception of rheumatoid nodule
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to rheumatoid arthritis
* History of cancer in the last 5 years, other than nonmelanoma skin cell cancer cured by local resection or carcinoma in situ. Existing nonmelanoma skin cell cancers should have been removed, the lesion site healed, and residual cancer ruled out prior to administration of study medication
* Clinically significant abuse of alcohol or drugs
* Evidence of active or latent bacterial or viral infections at the time of potential enrollment
* Herpes zoster or cytomegalovirus infection that resolved less than 2 months before the informed consent document was signed
* For participants at risk for tuberculosis (TB):

  * A history of active (TB) within the last 3 years, even if treated
  * Latent TB that was not successfully treated ≥4 weeks
  * Current clinical, radiographic, or laboratory evidence of active TB.
* Participants who have received live vaccines within 3 months of the anticipated first dose of study medication
* Participants with positive test results for hepatitis B surface antigen or hepatitis C antibody, with hepatitis C virus detected with polymerase chain reaction or recombinant immunoblot assay.
* Participants with hemoglobin level <8.5 g/dL or white blood cell count< 3000/mm^3 or platelet count <100,000/mm^3 or serum creatinin level >2*the upper limit of normal (ULN) or serum alanine transaminase level or aspartate aminotransferase level >2*ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- Local Institution, Glostrup Municipality, Denmark
- France (4):
  - Local Institution, Bois-Guillaume
  - Local Institution, Boulogne
  - Local Institution, Échirolles
  - Local Institution, Nice
- Local Institution, München, Germany
- Local Institution, Budapest, Hungary
- Italy (5):
  - Local Institution, Jesi (Ancona)
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Siena
  - Local Institution, Verona
- Norway (2):
  - Local Institution, Oslo
  - Local Institution, Trondheim
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Local Institution, Leeds, North Yorkshire, United Kingdom

REFERENCES:
- [Derived] D'Agostino MA, Boers M, Wakefield RJ, Berner Hammer H, Vittecoq O, Filippou G, Balint P, Moller I, Iagnocco A, Naredo E, Ostergaard M, Gaillez C, Le Bars M. Exploring a new ultrasound score as a clinical predictive tool in patients with rheumatoid arthritis starting abatacept: results from the APPRAISE study. RMD Open. 2016 May 5;2(1):e000237. doi: 10.1136/rmdopen-2015-000237. eCollection 2016. PMID 27175297
- [Derived] Golinski ML, Vandhuick T, Derambure C, Freret M, Lecuyer M, Guillou C, Hiron M, Boyer O, Le Loet X, Vittecoq O, Lequerre T. Dysregulation of RasGRP1 in rheumatoid arthritis and modulation of RasGRP3 as a biomarker of TNFalpha inhibitors. Arthritis Res Ther. 2015 Dec 26;17:382. doi: 10.1186/s13075-015-0894-9. PMID 26714738
- [Derived] D'Agostino MA, Wakefield RJ, Berner-Hammer H, Vittecoq O, Filippou G, Balint P, Moller I, Iagnocco A, Naredo E, Ostergaard M, Boers M, Gaillez C, Van Holder K, Le Bars M; OMERACT-EULAR-Ultrasound Task Force. Value of ultrasonography as a marker of early response to abatacept in patients with rheumatoid arthritis and an inadequate response to methotrexate: results from the APPRAISE study. Ann Rheum Dis. 2016 Oct;75(10):1763-9. doi: 10.1136/annrheumdis-2015-207709. Epub 2015 Nov 20. PMID 26590174
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 164 participants were screened; 104 were enrolled in the study and received open-label treatment with abatacept.
Groups:
- Abatacept, 10 mg/kg: All participants received abatacept by intravenous infusion at a fixed-dose approximating 10 mg/kg on Days 1, 15, 29, 57, 85, 113, 141, and 169 in addition to oral methotrexate. Abatacept dose was based on body weight at screening.
Period: Overall Study
Arm/Group | Abatacept, 10 mg/kg
Started | 104
Completed | 89
Not Completed | 15
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 3
Not completed — No longer met study criteria | 2
Not completed — Missed visit due to family reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 104
Age Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 101
  Other | 1
Tender joint count [Mean (Standard Deviation); unit: Joints] | 19.5 (12.5)
Duration of rheumatoid arthritis [Mean (Standard Deviation); unit: Years] | 7.3 (9.1)
Swollen joint count [Mean (Standard Deviation); unit: Joints] | 13.0 (7.6)
DAS 28-CRP score [Mean (Standard Deviation); unit: Units on a scale] — DAS28-CRP=Disease Activity Score 28 using C-Reactive Protein. The DAS28-CRP is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). These measures are then fed into a complex mathematical formula to produce the overall DAS (greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
  Units on a scale | 5.2888 (1.105)
Global PDUS (MCP 2-5) score (n=96) [Mean (Standard Deviation); unit: Units on a scale] — Power Doppler ultrasonography (PDUS) assessed synovial inflammation of metacarpophalangeal (MCP) joints (2-5) in both hands. Total PDUS score=sum of joints measured. Grade (Gr) 0, or normal=normal joint (no synovial hypertrophy(SH), no Doppler signal [[DS]); Gr 1 or minimal (min)=min synovitis (min SH with ≤Gr 1 Gr 2 or no DS); moderate (mod)=mod synovitis (mod SH with ≤Gr 2 Doppler signal or min SH and Gr 2 DS); Gr 3 or severe=severe synovitis (severe SH with ≤Gr 3 DS or min or mod SH and Gr 3 DS). Total possible score range: 8 to 24 (8*1, 8*3) for 2 hands. Higher grade=more severe disease.
  Units on a scale | 12.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Global Power Doppler Ultrasonography (PDUS) Score Assessing the Metacarpophalangeal (MCP) 2-5 Joints of Both Hands (LOCF Analysis)
Description: LOCF=last observation carried forward. PDUS assessed the degree of synovial inflammation of the MCP joints (2nd to 5th) of both hands and was performed at approximately the same time of day for each participant. Total PDUS scores are independent of the presence and grade of joint effusion and are evaluated as follows: Grade 0 or normal=normal joint (no synovial hypertrophy, no Doppler signal); Grade 1 or minimal=minimal synovitis (minimal synovial hypertrophy, with ≤Grade 1 Doppler signal); Grade 2 or moderate=moderate synovitis (moderate synovial hypertrophy with ≤Grade 2 Doppler signal or minimal synovial hypertrophy and Grade 2 Doppler signal; Grade 3 or severe=severe synovitis (severe synovial hypertrophy with ≤Grade 3 Doppler signal or minimal or moderate synovial hypertrophy and Grade 3 Doppler signal). Each joint is rated 1 to 3, for a total possible score ranging from 8 to 24 (8*1, 8*3) for 2 hands. Higher grade/score=more severe disease. Change=score Day x - baseline score.
Time Frame: Baseline to Days 7, 15, 29, 43, 57, 85, 113, 141, and 169
Population: All participants who received at least 1 infusion of study drug and who had baseline and at least 1 postbaseline efficacy measurements available. Excludes 8 participants with PDUS values from 1 site that experienced technical and quality issues with PDUS scoring and compliance.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 96
Units on a scale
  Day 7 (n=86) | -0.7 (0.282) [-1.2 to -0.1]
  Day 15 (n=94) | -1.3 (0.308) [-2.0 to -0.7]
  Day 29 (n=95) | -2.4 (0.383) [-3.2 to -1.7]
  Day 43 (n=95) | -2.9 (0.384) [-3.7 to -2.1]
  Day 57 (n=95) | -3.2 (0.393) [-4.0 to -2.4]
  Day 85 (n=95) | -3.8 (0.454) [-4.7 to -2.9]
  Day 113 (n=95) | -4.5 (0.472) [-5.4 to -3.5]
  Day 141 (n=95) | -4.8 (0.492) [-5.8 to -3.8]
  Day 169 (n=95) | -4.8 (0.473) [-5.8 to -3.9]
Statistical Analysis 1: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.2 to -0.1], Standard Error of Mean 0.282 — Day 7
Statistical Analysis 2: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.0 to -0.7], Standard Error of Mean 0.308 — Day 15
Statistical Analysis 3: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.2 to -1.7], Standard Error of Mean 0.383 — Day 29
Statistical Analysis 4: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-3.7 to -2.1], Standard Error of Mean 0.384 — Day 43
Statistical Analysis 5: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-4.0 to -2.4], Standard Error of Mean 0.393 — Day 57
Statistical Analysis 6: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-4.7 to -2.9], Standard Error of Mean 0.454 — Day 85
Statistical Analysis 7: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-5.4 to -3.5], Standard Error of Mean 0.472 — Day 113
Statistical Analysis 8: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-5.8 to -3.8], Standard Error of Mean 0.492 — Day 141
Statistical Analysis 9: Comparison: Abatacept, 10 mg/kg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-5.8 to -3.9], Standard Error of Mean 0.473 — Day 169

2. Secondary Outcome: Mean Change From Baseline in Global PDUS MCP 2-5 Component Scores Over Time (LOCF Analysis)
Description: PDUS=power Doppler ultrasonography; MCP=metacarpophalangeal; LOCF=last observation carried forward. PDUS was used to assess the degree of synovial inflammation of the MCP joints (2nd to 5th) of both hands and was performed at approximately the same time of day for each participant. PDUS scores are independent of the presence and grade of joint effusion and are evaluated as follows: Grade 0 or normal=normal joint (no synovial hypertrophy, no Doppler signal); Grade 1 or minimal=minimal synovitis (minimal synovial hypertrophy, with ≤Grade 1 Doppler signal); Grade 2 or moderate=moderate synovitis (moderate synovial hypertrophy with ≤Grade 2 Doppler signal or minimal synovial hypertrophy and grade 2 Doppler signal); Grade 3 or severe=severe synovitis (severe synovial hypertrophy with ≤ Grade 3 Doppler signal or minimal or 1-3, for a total possible score ranging from 8 to 24 (8*1, 8*3) for the 2 hands. Higher grade/score=more severe disease. Change=score Day X-baseline score.
Time Frame: Days 7, 15, 29, and 169
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 96
Units on a scale
  Synovial hypertrophy (n=86): Day 7 | -0.6 (0.297)
  Synovial hypertrophy (n=94): Day 15 | -1.0 (0.306)
  Synovial hypertrophy (n=95): Day 29 | -2.1 (0.377)
  Synovial hypertrophy (n=95): Day 169 | -4.5 (0.449)
  Doppler signal: Day 7 (n=86) | -0.9 (0.305)
  Doppler signal: Day 15 (n=94) | -1.9 (0.296)
  Doppler signal: Day 29 (n=95) | -2.2 (0.350)
  Doppler signal: Day 169 (n=95) | -4.8 (0.457)
  Joint effusion: Day 7 (n=86) | 0.1 (0.237)
  Joint effusion: Day 15 (n=94) | 0.1 (0.243)
  Joint effusion: Day 29 (n=95) | -0.8 (0.294)
  Joint effusion: Day 169 (n=95) | -1.9 (0.351)

3. Primary Outcome: Earliest Time Point at Which Improvement of Core Component of the Global PDUS in the MCP (2-5) Joints of Both Hands Was Assessed
Description: MCP=metacarpophalangeal; PDUS=power Doppler ultrasonography. Time point at which early signs of Global PDUS improvement were observed=earliest time point for which 0 was not included in the 95% confidence interval for the mean changes from baseline in Global PDUS (MCP 2-5) score at that and all later time points. Total PDUS scores are independent of the presence and grade of joint effusion: Grade (Gr) 0 or normal=normal joint (no synovial hypertrophy [SH], no Doppler signal); Gr 1 or minimal=minimal synovitis (minimal SH, with ≤Gr 1 Doppler signal); Gr 2 or moderate=moderate synovitis (moderate SH, with ≤Gr 2 Doppler signal or minimal SH and grade 2 Doppler signal); Gr 3 or severe=severe synovitis (severe SH with ≤Gr 3 Doppler signal or minimal or moderate SH and Gr 3 Doppler signal). Each joint is rated 1 to 3, for a total possible score ranging from 8 to 24 (8*1, 8*3) for the 2 hands. Higher Gr/score=more severe disease.
Time Frame: Baseline to Days 7, 15, 29, 43, 57, 85, 113, 141, and 169
Population: as for outcome 1
Measure: Number; unit: Day
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 96
Day | 7 [-1.5 to -0.3]

4. Secondary Outcome: Number of Early (Days 7 to 113) Global PDUS MCP 2-5 Scores or Global PDUS Component MCP 2-5 Scores Associated With an Acceptable Predictability of Clinical Response at Day 169, As Assessed by DAS28-CRP
Description: MCP=metacarpophalangeal; PDUS=power Doppler ultrasonography; DAS=Disease Activity Score;CRP=C-reactive protein. Receiver Operator Characteristics (ROC) analysis assessed predicatability. ROC curve analyses performed; area under the curve of ≥0.7 was considered acceptable for prediction. Clinical response defined as: Clinically Meaningful Improvement=drop from baseline of ≥1.2 in DAS28-CRP; Remission=DAS28-CRP score <2.6; Low Disease Activity=≤3.2. PDUS scores: Grade (Gr) 0 or normal=normal joint (no synovial hypertrophy [SH], no Doppler signal); Gr 1 or minimal=minimal synovitis (minimal SH, with ≤Gr 1 Doppler signal); Gr 2 or moderate=moderate synovitis (moderate SH with ≤Gr 2 Doppler signal or minimal SH and Gr 2 Doppler signal); Gr 3 or severe=severe synovitis (severe SH with ≤Gr 3 Doppler signal or minimal or moderate SH and Gr 3 Doppler signal). Each joint rated 1-3, for a total possible score ranging from 8-24 (8*1, 8*3)for the 2 hands. Higher gr/score=more severe disease.
Time Frame: Days 1 to 169
Population: as for outcome 1
Measure: Number; unit: Scores
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 96
Scores
  Clinically meaningful improvement | 0
  Remission | 0
  Low disease activity | 0

5. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events(SAEs), Treatment-related SAEs, Discontinuations Due to SAEs, Adverse Events (AEs), Treatment-related AEs, Discontinuations Due to AEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Days 1 to 169 to 56 days following last infusion
Population: All participants who received at least 1 infusion of study drug.
Measure: Number; unit: Participants
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 104
Participants
  Deaths | 0
  SAEs | 6
  Treatment-related SAEs | 2
  Discontinuations due to SAEs | 1
  AEs | 62
  Treatment-related AEs | 22
  Discontinuations due to AEs | 6

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) of Interest
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Infusion reaction: acute=1 hour or less after start of dosing; periinfusional=24 hours or less after start of dosing.
Time Frame: Days 1 to 169 to 56 days following last infusion
Population: All participants who received at least 1 infusion of study drug.
Measure: Number; unit: Participants
Arm/Group | Abatacept, 10 mg/kg
Number analyzed (Participants) | 104
Participants
  Infections | 20
  Malignancy | 1
  Autoimmune disorders (prespecified) | 2
  Infusion reactions (prespecified): Acute | 4
  Infusion reactions (prespecified): Periinfusional | 10

ADVERSE EVENTS:
Arm/Group | Aba 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 6/104
Other Adverse Events (participants affected / at risk) | 15/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aba 10 mg/kg (N=104)
Atrial fibrillation (Cardiac disorders) | 1
Bursitis infective (Infections and infestations) | 1
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1
Dementia (Nervous system disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aba 10 mg/kg (N=104)
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Nasopharyngitis (Infections and infestations) | 7

LIMITATIONS AND CAVEATS:
Power Doppler ultrasonography values from 1 site (8 participants were excluded due to technical and quality issues with PDUS scoring and compliance issues.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.